CLINICAL TRIAL: NCT06846528
Title: An Open-label, Fixed Sequence Study in Healthy Participants to Assess the Pharmacokinetics of AZD2389 When Administered Alone and in Combination With Itraconazole
Brief Title: A Study to Investigate the Pharmacokinetics of AZD2389 When Administered Alone and in Combination With Itraconazole in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D7930C00005
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Healthy Participants
Keywords: Fibroblast Activation Protein inhibitor; Advanced hepatic fibrosis; Chronic liver disease
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AZD2389 and Itraconazole (Experimental): AZD2389 is dosed on days 1 and 6. Itraconazole is dosed on days 3,4,5,6,7, with the dose on day 6 coming after AZD2389.
  Interventions: Drug: AZD2389; Drug: Itraconazole

INTERVENTIONS:
Drug: AZD2389 — AZD2389 is administered orally
Drug: Itraconazole — Itraconazole is administered orally

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (PK) of AZD2389 when administered alone and in combination with itraconazole in healthy participants.

DETAILED DESCRIPTION:
This study will be an open-label, fixed sequence, Drug-Drug Interaction (DDI) study consisting of 3 periods.

The study will comprise:

* A screening period of maximum 28 days
* Period 1
* Period 2
* Period 3
* A Follow-up Visit 7 to 14 days after the last PK sample has been collected.

ELIGIBILITY:
Inclusion Criteria:

* All females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit.
* Females of non-childbearing potential must be postmenopausal for at least 12 months or have documentation of irreversible surgical sterilization.
* Sexually active fertile male participants with partners of childbearing potential must adhere to the contraception methods.
* Have a Body Mass Index (BMI) between 18 and 32 kg/m2 inclusive and weigh at least 50 kg.

Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study intervention.
* Abnormal laboratory values, clinically important abnormalities or abnormal vital signs
* Any positive result on screening for serum Hepatitis B surface antigen/antibody, Hepatitis C, or Human Immunodeficiency Virus.
* Current smokers (within 3 months prior to screening visit) or history of alcohol and drug abuse
* History of severe allergy or hypersensitivity
* Excessive intake of caffeine-containing drinks or food
* Use of drugs with enzyme inducing properties or use of any prescribed or nonprescribed medication including antacids, analgesics

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Maximum observed drug concentration (Cmax) of AZD2389 | Day 1 to Day 8
  To assess the effect of itraconazole on the Cmax of AZD2389.
Area under concentration-timecurve from time zero to infinity (AUCinf) of AZD2389 | Day 1 to Day 8
  To assess the effect of itraconazole on the AUCinf of AZD2389.
Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) of AZD2389 | Day 1 to Day 8
  To assess the effect of itraconazole on the AUClast of AZD2389.

SECONDARY OUTCOMES:
Apparent total body clearance (CL/F) of AZD2389 | Day 1 to Day 8
  To describe the plasma PK of AZD2389 when AZD2389 is administered alone or in combination with itraconazole
Apparent volume of distribution based on the terminal phase (Vz/F) of AZD2389 | Day 1 to Day 8
  To describe the plasma PK of AZD2389 when AZD2389 is administered alone or in combination with itraconazole
Terminal elimination half-life (t1/2λz) of AZD2389 | Day 1 to Day 8
  To describe the plasma PK of AZD2389 when AZD2389 is administered alone or in combination with itraconazole.
Time to reach maximum observed concentration (tmax) of AZD2389 | Day 1 to Day 8
  To describe the plasma PK of AZD2389 when AZD2389 is administered alone or in combination with itraconazole.
Ratio of Test treatment (AZD2389 + itraconazole) to Reference (AZD2389) based on Cmax (RCmax) of AZD2389 | Day 1 to Day 8
  To describe the plasma PK of AZD2389 when AZD2389 is administered alone or in combination with itraconazole.
Ratio of Test treatment (AZD2389 + itraconazole) to Reference (AZD2389) based on AUClast (RAUClast) of AZD2389 | Day 1 to Day 8
  To describe the plasma PK of AZD2389 when AZD2389 is administered alone or in combination with itraconazole.
Ratio of Test treatment (AZD2389 + itraconazole) to Reference (AZD2389) based on AUCinf (RAUCinf) of AZD2389 | Day 1 to Day 8
  To describe the plasma PK of AZD2389 when AZD2389 is administered alone or in combination with itraconazole.
Renal Clearance (CLR) of AZD2389 | Day 1 to Day 8
  To describe the plasma PK of AZD2389 when AZD2389 is administered alone or in combination with itraconazole.
Individual and cumulative amount of unchanged drug excreted into urine from time t1 to time t2 (Ae(t1-t2)) of AZD2389 | Day 1 to Day 8
  To describe the plasma PK of AZD2389 when AZD2389 is administered alone or in combination with itraconazole.
Individual and cumulative percentage of dose excreted unchanged in urine from time t1 to time t2 (fe(t1-t2)) of AZD2389 | Day 1 to Day 8
  To describe the plasma PK of AZD2389 when AZD2389 is administered alone or in combination with itraconazole.
Percent change from baseline in fibroblast activation protein (FAP) inhibition | Day 1 to Day 8
  To evaluate the pharmacodynamics (PD) of AZD2389 by assessment of inhibition of FAP activity in plasma after single oral dose of AZD2389 alone or in combination with itraconazole.
Number of participants with Adverse Events (AEs) | From Screening (Day -29 to Day -2) up to 8 weeks
  To assess the safety and tolerability of a single oral dose of AZD2389 alone or in combination with itraconazole in healthy participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Brooklyn, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure."Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environmentVivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/